CLINICAL TRIAL: NCT04261829
Title: Autologous Fat Transfer: Introduction of a Full Breast Reconstructive Method
Brief Title: AFT: Introduction of a Full Breast Reconstructive Method
Acronym: BREAST-II
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: NL72808.068.20
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer; Reconstructive Surgery; Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autologous Fat Transfer
  Interventions: Procedure: Autologous Fat Transfer

INTERVENTIONS:
Procedure: Autologous Fat Transfer — Female breast cancer patients who were surgically treated with mastectomy could opt for a full breast reconstruction with Autologous Fat Transfer in combination with external expansion.
  Other Names: Lipofilling

SUMMARY:
A multicentre prospective cohort study will monitor the efficacy and safety of Autologous Fat Transfer (AFT) with pre-expansion. AFT will be evaluated in terms of quality of life, aesthetic result, complications, oncological safety and cost-effectiveness. It follows the BREAST trial, the randomised controlled trial comparing AFT with implant-based reconstruction. In this study, patients all receive AFT.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age of 18 years and older
* History or in candidate for a mastectomy procedure in the near future
* Patients undergoing preventive mastectomy
* Patients' choice to undergo a breast reconstruction
* Wanting to participate in this study
* Patient is able to wear the external expansion device

Exclusion Criteria:

* Active smoker or a history of smoking 4 weeks prior to surgery
* Current substance abuse
* History of lidocaine allergy
* History of silicone allergy
* 4 weeks or less after chemotherapy
* History of radiation therapy in the breast region
* Oncological treatment includes radiotherapy after mastectomy
* Kidney disease
* Steroid dependent asthma (daily or weekly) or other diseases
* Immune-suppressed or compromised disease
* Uncontrolled diabetes
* BMI>30
* Large breast size (i.e. larger than cup C), unless the patient prefers reduction of the contralateral side towards Cup C
* Extra-capsular silicone leaking from the encapsulated implant from a previous breast reconstruction
* The treating plastic surgeon has strong doubts on the patient's treatment compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Breast cancer patients or women who, due to a gene mutation have a significantly high risk of developing breast cancer, decide to undergo profylactic mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Breast-related Quality of life | 2 years
  Measured by the BREAST-Q questionnaire (quality of life subdivision)

SECONDARY OUTCOMES:
Aesthetic result | 2 years
  The overall aesthetic result will be measured using 3D-photographs which will be assessed by a panel of independent plastisch surgeons, ex-breast cancer patients and healthy volunteers. In addition, the volume, shape and symmetry will be assessed by the patient using the BREAST-Q questionnaire (satisfaction with breasts subdivisions).
Complications | 2 years
  Measurement of short-term als well as mid-term complications associated with procedures as well as (serious) adverse events.
Oncological safety | 5 years
  Oncological follow-up will comply to the guidelines for breast cancer and will take place by a yearly consult with the oncological surgeon (including physical examination and mammography/ultrasound/MRI) for 5 years postoperatively. All (loco)regional and distant recurrences will be recorded.
Cost-effectiveness | 2 years
  Cost-effectiveness analysis to determine the intramural and socio-economic costs associated with the breast reconstruction treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Piatkowski de Grzymala, MD, MSc, Principal Investigator — Maastricht University Medical Center
Locations (8):
- Netherlands (8):
  - Maastricht University Medical Center+, Maastricht, Limburg
  - Viecuri Venlo, Venlo, Limburg
  - Amsterdam University Medical Center (VUMC), Amsterdam
  - Rijnstate, Arnhem
  - Alexander Monro, Bilthoven, Bilthoven
  - Amphia, Breda
  - Ziekenhuis groep Twente (ZGT), Hengelo
  - Medical Center Leeuwarden, Leeuwarden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Venne WBW, Goeree KS, Wederfoort JLM, Hommes JE, van Kuijk SMJ, Heuts EM, Piatkowski de Grzymala AA, Moues CM; BREAST-II trial investigators. Evaluation of the BREAST-II Trial for Total Breast Reconstruction Solely Using Autologous Fat Transfer: 1-Year Follow-Up. Plast Reconstr Surg. 2026 Jan 22. doi: 10.1097/PRS.0000000000012742. Online ahead of print. PMID 41568954
- [Derived] Rijkx M, Saelmans A, Hommes J, Brandts L, De Bruijn D, Piatkowski A, Heuts E; Breast Reconstruction With External Preexpansion & autologous Fat Transfer vs Standard Therapy (BREAST) Trial Investigators. The Learning Curve of Total Breast Reconstruction With Autologous Fat Transfer. Ann Plast Surg. 2024 Oct 1;93(4):516-526. doi: 10.1097/SAP.0000000000004036. Epub 2024 Jul 15. PMID 39016317